CLINICAL TRIAL: NCT03391765
Title: An Extension Study of ABBV-8E12 in Progressive Supranuclear Palsy (PSP)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was prematurely discontinued because the program for progressive supranuclear palsy was discontinued due to lack of efficacy.
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M15-563; 2017-001590-16 (EudraCT Number)
Record Dates: First submitted 2018-01-02; First posted 2018-01-05 (Actual); Results first posted 2021-02-03 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Progressive Supranuclear Palsy (PSP)
Keywords: Tauopathy; Steele-Richardson-Olszewski Syndrome; PSP
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Tauopathies | interventions — tilavonemab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg (Experimental): Intravenous (IV) infusions of 2000 mg ABBV-8E12 at Day 1 and Day 29, then every 28 days for up to 5 years; administered at 300 mg/15 mL and 1000 mg/10 mL strength. Placebo IV infusion was administered on Day 15 in Study M15-563 (to maintain the blind in Study M15-562).
  Interventions: Drug: ABBV-8E12; Drug: Placebo solution for IV infusion on Day 15
- M15-562 ABBV-8E12 4000 mg/M15-563 ABBV-8E12 4000 mg (Experimental): Intravenous (IV) infusions of 4000 mg ABBV-8E12 at Day 1 and Day 29, then every 28 days for up to 5 years; administered at 300 mg/15 mL and 1000 mg/10 mL strength. Placebo IV infusion was administered on Day 15 in Study M15-563 (to maintain the blind in Study M15-562).
  Interventions: Drug: ABBV-8E12; Drug: Placebo solution for IV infusion on Day 15
- M15-562 Placebo/M15-563 ABBV-8E12 2000 mg (Experimental): Intravenous (IV) infusions of 2000 mg ABBV-8E12 at Day 1, Day 15, and Day 29, then every 28 days for up to 5 years; administered at 300 mg/15 mL and 1000 mg/10 mL strength.
  Interventions: Drug: ABBV-8E12
- M15-562 Placebo/M15-563 ABBV-8E12 4000 mg (Experimental): Intravenous (IV) infusions of 4000 mg ABBV-8E12 at Day 1, Day 15, and Day 29, then every 28 days for up to 5 years; administered at 300 mg/15 mL and 1000 mg/10 mL strength.
  Interventions: Drug: ABBV-8E12

INTERVENTIONS:
Drug: ABBV-8E12 — Participants with 44-49 kg body weight (BW) had an intravenous infusion rate of 3.5 mL/min or 210 mL/hr; those with 50-58 kg BW, 4.0 mL/min or 240 mL/hr; and those with a BW >59 kg, 4.7 mL/min or 282 mL/hr.
  Other Names: Tilavonemab
Drug: Placebo solution for IV infusion on Day 15 — 0.9% NaCl injection/solution for infusion 500 mL; participants with 44-49 kg body weight (BW) had an intravenous infusion rate of 3.5 mL/min or 210 mL/hr; those with 50-58 kg BW, 4.0 mL/min or 240 mL/hr; and those with a BW >59 kg, 4.7 mL/min or 282 mL/hr.
  Arms: M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg; M15-562 ABBV-8E12 4000 mg/M15-563 ABBV-8E12 4000 mg

SUMMARY:
The purpose of this study was to assess the long-term safety and efficacy of ABBV-8E12 (tilavonemab) in participants with progressive supranuclear palsy (PSP).

DETAILED DESCRIPTION:
This study (M15-563) was a Phase 2, randomized, double-blind, multiple-dose, multicenter, long-term extension of NCT 02985879 (Study M15-562) in participants with progressive supranuclear palsy (PSP). Those who completed the 52-week Treatment Period in Study M15-562 and met all entry criteria were eligible for enrollment into this study. This study planned for a Treatment Period of up to 5 years and a post-treatment follow-up visit approximately 20 weeks after the last dose of study drug (including participants who prematurely discontinued treatment). All participants received ABBV-8E12 as follows: those who received placebo in Study M15-562 were randomized, in a 1:1 ratio, to either 2000 or 4000 mg; those who received ABBV-8E12 at a dose of either 2000 or 4000 mg in Study M15-562 continued on the same dose in this study.

This study was prematurely discontinued because the program for progressive supranuclear palsy was discontinued due to lack of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Participant completed the 52-week treatment period in Study M15-562 (NCT02985879)
* In the opinion of the investigator, the participant was compliant during participation in Study M15-562 (NCT02985879)
* Participant has an identified, reliable, study partner (e.g., caregiver, family member, social worker, or friend)

Exclusion Criteria:

* Participants who weigh less than 44 kg (97 lbs) at the time of study entry
* Any contraindication or inability to tolerate brain magnetic resonance imaging (MRI)
* Participant has any significant change in his/her medical condition that could interfere with the subject's participation in the study, could place the subject at increased risk, or could confound interpretation of study results
* More than 8 weeks have elapsed since the participant received his/her last dose of study drug in Study M15-562 (NCT02985879)
* Participant is considered by the investigator, for any reason, to be an unsuitable candidate to receive ABBV-8E12 or the participant is considered by the investigator to be unable or unlikely to comply with the dosing schedule or study evaluations

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2019-12-13 (Actual); Study Completion 2019-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (42):
- United States (24):
  - Univ Alabama-Birmingham /ID# 165522, Birmingham, Alabama
  - Mayo Clinic Arizona /ID# 165521, Phoenix, Arizona
  - Cedars-Sinai Medical Center /ID# 165567, Beverly Hills, California
  - Usc /Id# 165529, Los Angeles, California
  - University of California, Los Angeles /ID# 165669, Los Angeles, California
  - University of California, San /ID# 165560, San Diego, California
  - Univ California, San Francisco /ID# 165553, San Francisco, California
  - Rocky Mountain Movement Disorders Center /ID# 165559, Englewood, Colorado
  - UF Center for Movement Disorde /ID# 165561, Gainesville, Florida
  - Mayo Clinic /ID# 165554, Jacksonville, Florida
  - University of South Florida /ID# 165556, Tampa, Florida
  - Augusta University Medical Center /ID# 165562, Augusta, Georgia
  - Rush University Medical Center /ID# 165527, Chicago, Illinois
  - University of Chicago Medical /ID# 165555, Chicago, Illinois
  - Indiana University /ID# 165519, Indianapolis, Indiana
  - University of Kentucky Chandler Medical Center /ID# 165566, Lexington, Kentucky
  - Mayo Clinic - Rochester /ID# 165518, Rochester, Minnesota
  - Cleveland Clinic Lou Ruvo Cent /ID# 165538, Las Vegas, Nevada
  - Rutgers Robert Wood Johnson /ID# 165526, New Brunswick, New Jersey
  - Columbia Univ Medical Center /ID# 165528, New York, New York
  - Cleveland Clinic Main Campus /ID# 165537, Cleveland, Ohio
  - Vanderbilt Univ Med Ctr /ID# 165520, Nashville, Tennessee
  - Kerwin Research Center /ID# 206872, Dallas, Texas
  - McGovern Medical School /ID# 165565, Houston, Texas
- Australia (3):
  - Q-Pharm Pty Limited /ID# 165452, Herston, Queensland
  - Royal Adelaide Hospital /ID# 165451, Adelaide, South Australia
  - Alfred Hospital /ID# 165454, Melbourne, Victoria
- Canada (4):
  - University of Calgary /ID# 165667, Calgary, Alberta
  - Toronto Western Hospital /ID# 165462, Toronto, Ontario
  - CHUM - Notre-Dame Hospital /ID# 165461, Montreal, Quebec
  - Montreal Neurological Institut /ID# 165546, Montreal, Quebec
- Italy (5):
  - Policlinico Agostino Gemelli /ID# 165536, Rome, Lazio
  - University of Catanzaro /ID# 170214, Catanzaro
  - Istituto Neuro Mediterraneo IR /ID# 165533, Pozzilli
  - A.O. Santa Maria /ID# 165535, Terni
  - IRCCS San Camillo /ID# 201229, Venice
- Japan (6):
  - National Hospital Organization Higashinagoya National Hospital /ID# 208786, Nagoya, Aichi-ken
  - National Hospital Organization Asahikawa Medical Center /ID# 208818, Asahikawa, Hokkaido
  - National Hospital Organization Utano National Hospital /ID# 208780, Kyoto, Kyoto
  - NHO Sendai Nishitaga National Hospital /ID# 209014, Sendai, Miyagi
  - Osaka University Hospital /ID# 208787, Suita-shi, Osaka
  - National Center of Neurology and Psychiatry /ID# 208820, Kodaira, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants
Period: Overall Study
Arm/Group | M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg | M15-562 ABBV-8E12 4000 mg/M15-563 ABBV-8E12 4000 mg | M15-562 Placebo/M15-563 ABBV-8E12 2000 mg | M15-562 Placebo/M15-563 ABBV-8E12 4000 mg
Started | 51 | 45 | 23 | 23
Completed | 0 | 0 | 0 | 0
Not Completed | 51 | 45 | 23 | 23
Not completed — Adverse Event | 2 | 0 | 0 | 2
Not completed — Withdrew consent | 5 | 7 | 2 | 5
Not completed — Other, not specified | 44 | 38 | 21 | 16

BASELINE CHARACTERISTICS:
Population: Stand-Alone Dataset: data from Study M15-563 only, regardless of the treatment received in Study M15-562. Baseline is the last observation on or before the first dose of ABBV-8E12 in Study M15-563. If no baseline was recorded in Study M15-563, the last value in Study M15-562 was used as baseline.
Groups:
- Total: Total of all reporting groups
Arm/Group | M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg | M15-562 ABBV-8E12 4000 mg/M15-563 ABBV-8E12 4000 mg | M15-562 Placebo/M15-563 ABBV-8E12 2000 mg | M15-562 Placebo/M15-563 ABBV-8E12 4000 mg | Total
Number analyzed (Participants) | 51 | 45 | 23 | 23 | 142
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (6.05) | 70.9 (6.58) | 68.8 (5.81) | 68.8 (5.78) | 69.9 (6.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 22 | 12 | 8 | 56
  Male | 37 | 23 | 11 | 15 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 47 | 42 | 22 | 22 | 133
  Black or African American | 2 | 1 | 0 | 0 | 3
  Asian | 1 | 2 | 1 | 1 | 5
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Multiple | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Progressive Supranuclear Palsy Rating Scale (PSPRS) Total Score From Baseline to Week 52
Description: The PSPRS consists of 28 items grouped in six domains: daily activities (by history); behavior; bulbar; ocular motor; limb motor; and gait/midline. Items are scored on a 0 to 4 scale, except for six items that are scored on a 0 to 2 scale, with the total score ranging from 0 to 100. Higher scores indicate more severe disability or movement abnormality. Positive values indicate worsening from baseline.
Time Frame: Baseline, Week 52
Population: ITT dataset: all participants who received any dose of study drug in Study M15-563 and those with available data at baseline and at Week 52
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg | M15-562 ABBV-8E12 4000 mg/M15-563 ABBV-8E12 4000 mg | M15-562 Placebo/M15-563 ABBV-8E12 2000 mg | M15-562 Placebo/M15-563 ABBV-8E12 4000 mg
Number analyzed (Participants) | 9 | 6 | 7 | 6
units on a scale | 14.4 (7.73) | 2.3 (11.99) | 13.1 (6.87) | 4.2 (6.40)

2. Secondary Outcome: Mean Change From Baseline to Week 52 in Unified Parkinson's Disease Rating Scale (UPDRS) Part II (Activities of Daily Living)
Description: The Unified Parkinson's Disease Rating Scale (UPDRS) is an Investigator-used rating tool to follow the longitudinal course of Parkinson's disease. The Part II score is the sum of the answers to the 13 questions related to Activities of Daily Living, and ranges from 0-52. Higher scores are associated with more disability. Positive values indicate worsening from baseline.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg | M15-562 ABBV-8E12 4000 mg/M15-563 ABBV-8E12 4000 mg | M15-562 Placebo/M15-563 ABBV-8E12 2000 mg | M15-562 Placebo/M15-563 ABBV-8E12 4000 mg
Number analyzed (Participants) | 9 | 6 | 7 | 6
units on a scale | 6.9 (4.37) | 3.2 (5.27) | 5.6 (5.68) | 7.3 (6.28)

3. Secondary Outcome: Change in Clinical Global Impression of Severity (CGI-C) Score From Baseline to Week 52
Description: The Clinical Global Impression of Change (CGI-C) score is a clinician's rating scale for assessing Global Improvement of Change. The CGI-C rates improvement by 7 categories: very much improved (1), much improved (2), minimally improved (3), no change (4), minimally worse (5), much worse (6), very much worse (7). The CGI-C score ranges from 1 to 7, with lower scores indicating improvement.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg | M15-562 ABBV-8E12 4000 mg/M15-563 ABBV-8E12 4000 mg | M15-562 Placebo/M15-563 ABBV-8E12 2000 mg | M15-562 Placebo/M15-563 ABBV-8E12 4000 mg
Number analyzed (Participants) | 50 | 42 | 22 | 23
units on a scale
  Baseline of M15-563 | 5.0 (0.89) | 4.8 (0.92) | 4.9 (0.92) | 5.0 (0.91)
  Week 52 of M15-563: number analyzed (Participants) | 8 | 6 | 7 | 5
  Week 52 of M15-563 | 5.1 (0.64) | 5.2 (0.98) | 5.9 (0.90) | 5.4 (1.14)

4. Secondary Outcome: Mean Change From Baseline to Week 52 in Schwab and England Activities of Daily Living Scale (SEADL)
Description: The Schwab and England Activities of Daily Living (SEADL) scale consists of ten items intended to evaluate the daily life activities of a participant. The SEADL is composed of two sections: the first is a self-reported questionnaire in which participants grade their own daily life activities, such as dressing, using the toilet, resting, eating, and social activities (subjective assessment), and the second is an assessment of motor functions, such as postural balance, speaking, rigidity, and tremors, conducted by a clinician (objective assessment). It is a percentage scale divided into deciles, and the results are reported between 0% (bedridden) and 100% (healthy). Negative values indicate worsening from baseline.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg | M15-562 ABBV-8E12 4000 mg/M15-563 ABBV-8E12 4000 mg | M15-562 Placebo/M15-563 ABBV-8E12 2000 mg | M15-562 Placebo/M15-563 ABBV-8E12 4000 mg
Number analyzed (Participants) | 9 | 6 | 7 | 5
units on a scale | -13.3 (14.14) | -13.3 (12.11) | -10.0 (14.14) | -18.0 (13.04)

5. Secondary Outcome: Mean Change From Baseline to Week 52 in Clinical Global Impression of Severity (CGI-S) Score
Description: The CGI-S is a clinician's rating of disease severity. The CGI-S rates severity of illness on a 7-point scale, using a range of responses from 1 (normal) through 7 (the most severely ill). This rating is based upon observed and reported symptoms, behavior, and function in the past 7 days. Positive values indicate worsening from baseline.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg | M15-562 ABBV-8E12 4000 mg/M15-563 ABBV-8E12 4000 mg | M15-562 Placebo/M15-563 ABBV-8E12 2000 mg | M15-562 Placebo/M15-563 ABBV-8E12 4000 mg
Number analyzed (Participants) | 8 | 6 | 7 | 5
units on a scale | 0.6 (0.52) | 1.3 (0.82) | 1.3 (0.49) | 0.6 (1.82)

6. Secondary Outcome: Patient Global Impression of Change Score (PGI-C) Score From Baseline to Week 52
Description: The PGI-C is a participant's rating of the change in their PSP-related symptoms since initiation of study drug. Participants rated their change in status using the following 7-point scale: 1 = Very much improved; 2 = Much improved; 3 = Minimally improved; 4 = No change; 5 = Minimally worse; 6 = Much worse; 7 = Very much worse.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg | M15-562 ABBV-8E12 4000 mg/M15-563 ABBV-8E12 4000 mg | M15-562 Placebo/M15-563 ABBV-8E12 2000 mg | M15-562 Placebo/M15-563 ABBV-8E12 4000 mg
Number analyzed (Participants) | 48 | 43 | 23 | 23
units on a scale
  Baseline of M15-563 | 5.0 (1.03) | 5.1 (1.04) | 5.2 (1.30) | 5.3 (1.15)
  Week 52 of M15-563: number analyzed (Participants) | 9 | 6 | 7 | 6
  Week 52 of M15-563 | 4.9 (1.62) | 4.7 (1.51) | 5.4 (0.53) | 5.3 (1.37)

7. Secondary Outcome: Mean Change From Baseline to Week 52 in Progressive Supranuclear Palsy Staging System Score (PSP-SS) Score
Description: The Progressive Supranuclear Palsy Rating Scale (PSPRS) consists of 28 items grouped in six domains: daily activities (by history); behavior; bulbar; ocular motor; limb motor; and gait/midline. Items are scored on a 0 to 4 scale, except for four items that are scored on a 0 to 2 scale, with the total score ranging from 0 to 100. Higher scores indicate more severe disability or movement abnormality. The PSP-SS score is a composite of the dysphagia and gait items from the PSPRS. Positive values indicate worsening from baseline.
Time Frame: Baseline, Week 52
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg | M15-562 ABBV-8E12 4000 mg/M15-563 ABBV-8E12 4000 mg | M15-562 Placebo/M15-563 ABBV-8E12 2000 mg | M15-562 Placebo/M15-563 ABBV-8E12 4000 mg
Number analyzed (Participants) | 9 | 6 | 7 | 6
units on a scale | 2.4 (1.74) | -0.2 (2.23) | 2.0 (2.83) | 1.0 (2.10)

8. Secondary Outcome: Time to Loss of Ability to Walk Independently as Measured by Progressive Supranuclear Palsy Rating Scale (PSPRS) Item 26
Description: The PSPRS consists of 28 items grouped in six domains: daily activities (by history); behavior; bulbar; ocular motor; limb motor; and gait/midline. Items are scored on a 0 to 4 scale, except for four items that are scored on a 0 to 2 scale, with the total score ranging from 0 to 100. Higher scores indicate more severe disability or movement abnormality. Item 26 pertains to gait, scored as either 0 (normal); 1 (slightly wide-based or irregular or slight pulsion on turns); 2 (must walk slowly or occasionally use walls or helper to avoid falling, especially on turns); 3 (must use assistance all or almost all the time); or 4 (unable to walk, even with walker; may be able to transfer).
Time Frame: From Baseline to Week 52
Population: ITT dataset: all participants who received any dose of study drug in Study M15-563 and those with available data
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg | M15-562 ABBV-8E12 4000 mg/M15-563 ABBV-8E12 4000 mg | M15-562 Placebo/M15-563 ABBV-8E12 2000 mg | M15-562 Placebo/M15-563 ABBV-8E12 4000 mg
Number analyzed (Participants) | 51 | 45 | 23 | 23
days | 84.0 [29.0 to 86.0] | 85.0 [84.0 to 91.0] | 85.0 [42.0 to 91.0] | 84.0 [64.0 to 86.0]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from the first dose of study drug until 20 weeks following discontinuation of study drug administration have elapsed (approximately 5 half-lives), up to 98 weeks. In addition, serious adverse events and protocol-related nonserious adverse events were collected from the time the participant signed the study-specific informed consent.
Description: TEAEs and SAEs are defined as any AE or SAE with onset or worsening reported by a participant from the time that the first dose of study is administered until 20 weeks (approximately 5 half-lives) have elapsed following discontinuation of study drug. TEAEs were collected whether elicited or spontaneously reported by the participant.
Groups:
- M15-562 ABBV-8E12 4000 mg /M15-563 ABBV-8E12 4000 mg: Intravenous (IV) infusions of 4000 mg ABBV-8E12 at Day 1 and Day 29, then every 28 days for up to 5 years; administered at 300 mg/15 mL and 1000 mg/10 mL strength. Placebo IV infusion was administered on Day 15 in Study M15-563 (to maintain the blind in Study M15-562).
Arm/Group | M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg | M15-562 ABBV-8E12 4000 mg /M15-563 ABBV-8E12 4000 mg | M15-562 Placebo/M15-563 ABBV-8E12 2000 mg | M15-562 Placebo/M15-563 ABBV-8E12 4000 mg
All-Cause Mortality (participants affected / at risk) | 5/51 | 5/45 | 1/23 | 2/23
Serious Adverse Events (participants affected / at risk) | 10/51 | 10/45 | 3/23 | 7/23
Other Adverse Events (participants affected / at risk) | 18/51 | 16/45 | 6/23 | 16/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg (N=51) | M15-562 ABBV-8E12 4000 mg /M15-563 ABBV-8E12 4000 mg (N=45) | M15-562 Placebo/M15-563 ABBV-8E12 2000 mg (N=23) | M15-562 Placebo/M15-563 ABBV-8E12 4000 mg (N=23)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COMPLICATION ASSOCIATED WITH DEVICE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEATH (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
KLEBSIELLA INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 3 (5) | 0 (0) | 0 (0) | 0 (0)
POST PROCEDURAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
RIB FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLORECTAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LYMPHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PARTIAL SEIZURES (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROGRESSIVE SUPRANUCLEAR PALSY (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
APNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | M15-562 ABBV-8E12 2000 mg/M15-563 ABBV-8E12 2000 mg (N=51) | M15-562 ABBV-8E12 4000 mg /M15-563 ABBV-8E12 4000 mg (N=45) | M15-562 Placebo/M15-563 ABBV-8E12 2000 mg (N=23) | M15-562 Placebo/M15-563 ABBV-8E12 4000 mg (N=23)
CONSTIPATION (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0) | 2 (2)
DYSPHAGIA (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 7 (11) | 7 (10) | 1 (1) | 2 (2)
CHEST INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CONTUSION (Injury, poisoning and procedural complications) | 2 (3) | 3 (4) | 1 (2) | 2 (5)
FALL (Injury, poisoning and procedural complications) | 9 (13) | 7 (9) | 2 (8) | 9 (20)
LIP INJURY (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
SKIN ABRASION (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 2 (2) | 3 (3)
SKIN LACERATION (Injury, poisoning and procedural complications) | 5 (5) | 3 (3) | 1 (4) | 6 (9)
WEIGHT DECREASED (Investigations) | 2 (2) | 0 (0) | 1 (2) | 3 (3)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3)
ANXIETY (Psychiatric disorders) | 0 (0) | 4 (4) | 2 (2) | 1 (1)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/65/NCT03391765/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/65/NCT03391765/SAP_001.pdf